CLINICAL TRIAL: NCT01463800
Title: Cardiac Rehabilitation in Patients With Complex Congenital Heart Disease: Improvement of Exercise Intolerance
Brief Title: Rehabilitation in Patients With Congenital Heart Disease
Acronym: CARE-GUCH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low inclusion rate
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CARE-GUCH
Record Dates: First submitted 2011-10-28; First posted 2011-11-02 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Heart Defects, Congenital
Keywords: Heart Defects, congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured Exercise training (Active Comparator): 12 weeks ambulatory low level exercise training
  Interventions: Behavioral: Structured exercise training
- Control group (No Intervention): No structured exercise training

INTERVENTIONS:
Behavioral: Structured exercise training — 12 weeks low level ambulatory structured exercise training
  Arms: Structured Exercise training

SUMMARY:
Exercise intolerance is a major burden for patients with complex congenital heart disease (CHD), significantly affecting their quality of life. Cardiopulmonary exercise testing provides a reliable tool both for assessing exercise capacity of CHD patients and for risk stratification and is becoming part of the routine clinical assessment of these patients. Exercise has an effect on the muscular, metabolic and circulatory systems. While exercise training has been widely studied in chronic heart failure, its efficacy in adults with CHD remain unknown. The investigators hypothesize that structured exercise training will improve exercise intolerance, in particular peak VO2. The aim of this multicenter, randomized study is to evaluate the impact of structured exercise training on exercise intolerance in patients with complex CHD.

DETAILED DESCRIPTION:
This is a randomized, prospective, multicenter, interventional study.

After study patients have given written consent they will be randomized either in the interventional group with a rehabilitation program or in the control group without rehabilitation program. Patients who are randomized in the control group are allowed to perform the rehabilitation program 12 months after randomisation. Patients in the interventional group will perform structured exercise training on 3 weekdays during a 12-weeks period. Training will be performed by ergometer and low-impact gymnastic and relaxation training.

All study participants have the following investigations at the beginning of the study and after 12 weeks:

* Cardiopulmonary exercise testing with spirometry
* 6-minute walk test
* Blood work: BNP, Creatinine, Sodium, Potassium, Urat, Cholesterol (HDL-L and LDL-L)
* Validated Heart failure questionnaires (SF-36 and Minnesota Living with heart failure questionnaire, German version for Basel, Zürich and Bern) All tests will be repeated as clinically indicated in a follow-up visit 12 months after baseline

Primary outcome is:

Comparison of peak VO2 at the end of rehabilitation between both groups.

Secondary outcomes are:

* Comparison of 6-min walk test, VE/VCO2 slope, anaerobic threshold and heart rate and blood pressure response after rehabilitation between both groups
* Changes of 6-min walk test, peak VO2, VE/VCO2 slope, anaerobic threshold and heart rate and blood pressure response at the end and 12 months after rehabilitation.
* Changes of quality-of-life assessed by validated heart failure questionnaire at the end and 12 months after rehabilitation and comparison between both groups.
* Changes of levels of brain-natriuretic peptide at the end and 12 months after rehabilitation.
* Adverse events during rehabilitation including new onset of arrhythmia, admission due to worsening heart failure or death.

The calculated sample size to reach a power of 0.80 is 83 patients in each arm. Patients with complex CHD and exercise intolerance are at increased risk for premature death and severe cardiac complications including arrhythmia needing treatment, heart failure and circulatory failure, pulmonary hemorrhage, pulmonary embolism and endocarditis. Hence, the likelihood of major adverse cardiac events during the study phase is considerably high. However, there is no evidence of functional worsening by low-level exercise. Smaller studies with patients with congenital heart disease and/or pulmonary hypertension did not report safety issues. Although sudden cardiac death is one of the leading modes of death in this population, it is extremely rare that sudden death occurs during exercise. Cardiac patients who are at specific risk for exercise-induced arrhythmia are not included into the study (i.e. patients with hypertrophic obstructive cardiomyopathy).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with complex CHD including cyanotic heart disease, subaortic right ventricle physiology, single ventricle physiology, Ebstein anomaly with ≥ moderate tricuspid regurgitation and patients with Tetralogy of Fallot (including those with pulmonary atresia of Fallot type or double-outlet right ventricle of Fallot type) and either residual free pulmonary regurgitation or left- or right ventricular systolic dysfunction (demonstrated by echocardiography or cardiac MRI).
2. Peak VO2 < 85% of predicted (standardized for age, gender, weight and height) obtained by cardiopulmonary exercise testing
3. Sedentary lifestyle (< 30 minutes of regular exercise per week)

Exclusion Criteria:

1. Patients with dyspnea New York Heart Association (NYHA) class IV.
2. Severe left ventricular outflow tract obstruction.
3. Unstable angina or recent myocardial infarction (<12 months).
4. Uncontrolled ventricular arrhythmia.
5. Recent intervention (<12 months)
6. Life expectancy <12 months
7. No consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-05; Primary Completion 2016-05 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
peak VO2 | 12 weeks
  Comparison between both groups

SECONDARY OUTCOMES:
6 minute walk test | 12 weeks
  between both groups and within groups
VE/VCO2 | 12 weeks
  Comparison between groups and within groups
heart rate response | 12 weeks
  Difference between peak heart rate and resting heart rate Comparison between groups and within groups
QoL | 12 weeks
  Comparison between groups and within groups Minnesota Heart failure Score and SF 36
BNP | 12 weeks
  Comparison between groups and within groups
Adverse events | 12 weeks
  cardiac related adverse events including cardiac death
peak VO2 | 12 months
  Comparison between groups and within groups
VE/VCO2 | 12 months
  Comparison between groups and within groups
Heart rate response | 12 months
  Comparison between groups and within groups
6 minute walk test | 12 months
  Comparison between groups and within groups
QoL | 12 months
  Comparison between groups and within groups
BNP | 12 months
  Comparison between groups and within groups
Cardiac adverse events | 12 months
  Comparison between groups and within groups

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tobler, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (4):
- Virgen Macarena University Hospital, Seville, Spain
- Switzerland (3):
  - University Hospital Basel, Basel
  - Inselspital Bern, Bern
  - University Hospital Zurich, Zurich